CLINICAL TRIAL: NCT01476943
Title: Belatacept in Renal Transplantation: Patterns of Use Analysis Using the Collaborative Transplant Study (CTS)
Brief Title: Patterns of Use of Belatacept: Analysis of Data From the Collaborative Transplant Study
Acronym: CTS
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: IM103-077
Record Dates: First submitted 2011-11-08; First posted 2011-11-22 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Transplantation, Organ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient treated with Belatacept at the time of transplantation: Patients undergoing solid organ transplantation, whose transplant center participates in CTS and who are treated with Belatacept at the time of transplantation
- Patient treated with CNI at the time of transplantation: Patients undergoing solid organ transplantation, whose transplant center participates in CTS and who are treated with a Calcineurin inhibitor (CNI) based regimen at the time of transplantation

SUMMARY:
The primary purpose is to describe the pattern of Belatacept use at the time of transplant and up to three years post-transplantation for all Belatacept treated patients.

DETAILED DESCRIPTION:
Time Perspective: Prospective design, Retrospective data collection and analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients who received solid organ transplantation during study period in one of the transplant centers involved in CTS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing solid organ transplantation, whose transplant center participates in CTS and who are treated with Belatacept or a CNI based regimen at the time of transplantation
Sampling Method: Non-Probability Sample
Enrollment: 72392 (Actual)
Dates: Start 2012-03-31 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
The number and percent of belatacept users overall, by Epstein-Barr Virus (EBV) serostatus and by Cytomegalovirus (CMV) serostatus | At the time of transplantation
The number and percent of belatacept users overall, by Epstein-Barr Virus (EBV) serostatus and by CMV serostatus | 1 year post transplantation
The number and percent of belatacept users overall, by Epstein-Barr Virus (EBV) serostatus and by CMV serostatus | 2 year post transplantation
The number and percent of belatacept users overall, by Epstein-Barr Virus (EBV) serostatus and by CMV serostatus | 3 year post transplantation

SECONDARY OUTCOMES:
Extent of switches to or from Belatacept within three years post transplantation, and the temporal trend in switches post regulatory approval of Belatacept | At transplantation, 12 month, 24 month and 36 month post transplantation
Characteristics of Belatacept users vs. Calcineurin inhibitor (CNIs) users at transplantation | At the time of transplantation
Characteristics of those who switch to or from Belatacept vs. those who do not switch one year post-transplant | At transplantation and 12 month post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm